CLINICAL TRIAL: NCT07300540
Title: A Real-World Evidence Study Evaluating Oral Health Related Quality of Life With Use of a Calcium Sodium Phosphosilicate Anti-Sensitivity Dentifrice for Dentin Hypersensitivity Management
Brief Title: Real-World Study of a Calcium Sodium Phosphosilicate Anti-Sensitivity Toothpaste for Dentin Hypersensitivity Relief
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 400303
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Toothpastes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Toothpaste (Other): Participants will be instructed to brush their teeth twice daily and not more than three times per day using test toothpaste, for 24 weeks.
  Interventions: Other: Calcium sodium phosphosilicate (CSPS) Toothpaste

INTERVENTIONS:
Other: Calcium sodium phosphosilicate (CSPS) Toothpaste — A toothpaste containing 5% weight/weight (w/w) calcium sodium phosphosilicate.

SUMMARY:
The aim of this study is to evaluate the impact of a commercially available desensitizing dentifrice containing 5 percent (%) Calcium sodium phosphosilicate (CSPS) on oral health related quality of life (OHrQoL) in a DH (Dentin Hypersensitivity) population in a real-world setting.

DETAILED DESCRIPTION:
This will be a decentralized, prospective, 24-week, monadic design, open label, study in a DH population. The study will evaluate changes in OHrQoL in participants with self-reported DH symptoms. OHrQoL will be measured using a validated questionnaire, the Dentin Hypersensitivity Experience Questionnaire (DHEQ-48), completed by study participant. Sufficient numbers will be screened to enroll approximately 500 participants to ensure approximately 400 evaluable participants complete the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Participant who has provided consent indicating they have been informed of all pertinent aspects of the study.
* All genders who, at the time of screening, are aged 18 to 65.
* Participant who is able to independently complete all activities on their smart devices
* Participant who has tooth sensitivity (self-reported symptoms).

Exclusion Criteria:

* Participants whose tooth sensitivity could be caused by other factors or clinical pathology than DH, as self-reported on the screening questionnaire, which include:

  1. Participant who has been/is on multiple prescription medications to treat severe acid reflux on a regular basis or has had surgery for acid reflux.
  2. Participant with full or partial denture.
  3. Participant who has undergone treatment for periodontal or gum disease within 6 months of screening or is currently undergoing treatment for periodontal or gum disease.
  4. Participant who has been informed by a Dental Health Care Professional (DHCP) that they have active periodontitis.
  5. Participants who have been informed by a DHCP that they have active caries.
  6. Participant with any chronic and/or severe painful health condition which lead to regular use of pain relief medications (more than 3 days a week).
* Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in DHEQ Total Score at Week 24 | Baseline and Week 24
  The DHEQ is used to measure how DH affects participants quality of life. Section 2 has 34 questions in grouped into 5 domains (Restrictions, Adaptation, Social Impact, Emotional Impact, and Identity). Participants scored each question using a 7-point scale ranging from 1 to 7, where 1= strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score will be derived from the sum of scores across all domains and it ranges from 34 to 238. A lower score indicates a better quality of life regarding DH. Change from Baseline will be calculated by subtracting the Baseline score from the score at Week 24.

SECONDARY OUTCOMES:
Change From Baseline in DHEQ Restrictions Domain Score at Week 24 | Baseline and Week 24
  Restrictions domain of DHEQ evaluates 'the ways in which any sensations in teeth affects participants in their daily life'. It includes 4 questions, each will be scored using 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree, resulting in a total score ranging from 4 to 28. A lower score indicates that sensations have less effect on daily life. Changes from a baseline will be calculated by subtracting the baseline score from the score at Week 24.
Change From Baseline in DHEQ Adaptation Domain Score at Week 24 | Baseline and Week 24
  Adaptation domain of DHEQ evaluates 'the ways in which the sensations in teeth forces participants to change things in their daily life'; 'things they do in their daily life to avoid experiencing the sensations in their teeth'. It includes 12 questions, each will be scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranges from 12 to 84, where lower score indicates less effect of sensations on participant's daily life. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 24.
Change From Baseline in DHEQ Social Impact Domain Score at Week 24 | Baseline and Week 24
  Social Impact domain of DHEQ assesses how sensations affect participants in social situations. It includes 5 questions each will be scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score ranges from 5 to 35. A lower score indicates less effect of sensations on participant's social life. Change from baseline is calculated by subtracting the baseline score from score at Week 24.
Change From Baseline in DHEQ Emotional Impact Domain Score at Week 24 | Baseline and Week 24
  Emotional Impact Domain of DHEQ is used to assess the emotional impact of sensations in participant's teeth. It includes 8 questions each will be scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score ranges from 8 to 56, where lower score indicated less impact of sensations on participant's emotions. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 24.
Change From Baseline in DHEQ Identity Domain Score at Week 24 | Baseline and Week 24
  Identity Domain of DHEQ evaluated 'what the sensations in participant's teeth mean for them'. It includes 5 questions each will be scored using 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score ranges from 5 to 35, where lower score indicates less impact of sensations on participant's identity. Change from baseline is calculated by subtracting the baseline score from score at Week 24.
Change From Baseline in Impact on Everyday Life Score at Week 24 | Baseline and Week 24
  Impact on Everyday Life section of DHEQ includes 3 questions about participant's sensitive teeth and its impact on everyday life. Participants will score Q1 (how intense are the sensations?) on a scale of 1 (not at all intense) to 10 (worst imaginable); Q2 (how bothered are you by any sensations?) on a scale of 1 (not at all bothered) to 10 (extremely bothered); Q3 (how well can you tolerate sensations?) on a scale of 1 (can easily tolerate) to 10 (can't tolerate at all). The total score for each question ranges from 1 to 10; where lower scores indicate less intense, less bothersome and tolerable sensations. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 24.
Change From Baseline in Global Oral Health Score at Week 24 | Baseline and Week 24
  Global Oral Health is evaluated using a single question of DHEQ. Participants will rate the overall health of their mouth, teeth, and gums using a 6-point scale ranging from 1 to 6 where 1=excellent, 2=very good, 3=good, 4=fair, 5=poor, and 6=very poor. Lower score indicates better oral health. Change from baseline will be calculated by subtracting the baseline score from score at Week 24.
Change From Baseline in Effect on Life Overall Score at Week 24 | Baseline and Week 24
  Effect on life will be evaluated using 4 questions of DHEQ about how much the sensation in teeth affects participant's life overall. Participants will score each question on a 5-point scale ranging from 0 to 4 where 0=not at all, 1=a little, 2=somewhat; 3=quite a bit, and 4=very much. Thus, the total score ranges from 0 to 16, where lower score indicates less effect of sensations on participant's life overall. Change from Baseline will be calculated by subtracting the Baseline score from score at Week 24.
Change From Baseline in Impact on Everyday Life Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Impact on Everyday Life section of DHEQ includes 3 questions about participant's sensitive teeth and its impact on everyday life. Participants will score Q1 (how intense are the sensations?) on a scale of 1 (not at all intense) to 10 (worst imaginable); Q2 (how bothered are you by any sensations?) on a scale of 1 (not at all bothered) to 10 (extremely bothered); Q3 (how well can you tolerate sensations?) on a scale of 1 (can easily tolerate) to 10 (can't tolerate at all). The total score for each question ranges from 1 to 10; where lower scores indicate less intense, less bothersome and tolerable sensations. Change from Baseline will be calculated by subtracting the Baseline score from score at the indicated timepoints.
Change From Baseline in DHEQ Total Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  The DHEQ is used to measure how DH affects participants quality of life. Section 2 has 34 questions in grouped into 5 domains (Restrictions, Adaptation, Social Impact, Emotional Impact, and Identity). Participants scored each question using a 7-point scale ranging from 1 to 7, where 1= strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score will be derived from the sum of scores across all domains and it ranges from 34 to 238. A lower score indicates a better quality of life regarding DH. Change from Baseline will be calculated by subtracting the Baseline score from the score at the indicated timepoints.
Change From Baseline in DHEQ Restrictions Domain Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Restrictions domain of DHEQ evaluates 'the ways in which any sensations in teeth affects participants in their daily life'. It includes 4 questions, each will be scored using 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree, resulting in a total score ranging from 4 to 28. A lower score indicates that sensations have less effect on daily life. Changes from a baseline will be calculated by subtracting the baseline score from the score at the indicated timepoints.
Change From Baseline in DHEQ Adaptation Domain Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Adaptation domain of DHEQ evaluates 'the ways in which the sensations in teeth forces participants to change things in their daily life'; 'things they do in their daily life to avoid experiencing the sensations in their teeth'. It includes 12 questions, each will be scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. Thus, the total score ranges from 12 to 84, where lower score indicates less effect of sensations on participant's daily life. Change from Baseline will be calculated by subtracting the Baseline score from score at the indicated timepoints.
Change From Baseline in DHEQ Social Impact Domain Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Social Impact domain of DHEQ assesses how sensations affect participants in social situations. It includes 5 questions each will be scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score ranges from 5 to 35. A lower score indicates less effect of sensations on participant's social life. Change from baseline is calculated by subtracting the baseline score from score at the indicated timepoints.
Change From Baseline in DHEQ Emotional Impact Domain Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Emotional Impact Domain of DHEQ is used to assess the emotional impact of sensations in participant's teeth. It includes 8 questions each will be scored using a 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score ranges from 8 to 56, where lower score indicated less impact of sensations on participant's emotions. Change from Baseline will be calculated by subtracting the Baseline score from score at the indicated timepoints.
Change From Baseline in DHEQ Identity Domain Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Identity Domain of DHEQ evaluated 'what the sensations in participant's teeth mean for them'. It includes 5 questions each will be scored using 7-point scale ranging from 1 to 7 where 1=strongly disagree, 2=disagree, 3=disagree a little, 4=neither agree nor disagree, 5=agree a little, 6=agree, and 7=strongly agree. The total score ranges from 5 to 35, where lower score indicates less impact of sensations on participant's identity. Change from baseline is calculated by subtracting the baseline score from score at the indicated timepoints.
Change From Baseline in Global Oral Health Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Global Oral Health is evaluated using a single question of DHEQ. Participants will rate the overall health of their mouth, teeth, and gums using a 6-point scale ranging from 1 to 6 where 1=excellent, 2=very good, 3=good, 4=fair, 5=poor, and 6=very poor. Lower score indicates better oral health. Change from baseline will be calculated by subtracting the baseline score from score at the indicated timepoints.
Change From Baseline in Effect on Life Overall Score at Weeks 4, 8, 12, 16, and 20 | Baseline and Weeks 4, 8, 12, 16, 20
  Effect on life will be evaluated using 4 questions of DHEQ about how much the sensation in teeth affects participant's life overall. Participants will score each question on a 5-point scale ranging from 0 to 4 where 0=not at all, 1=a little, 2=somewhat; 3=quite a bit, and 4=very much. Thus, the total score ranges from 0 to 16, where lower score indicates less effect of sensations on participant's life overall. Change from Baseline will be calculated by subtracting the Baseline score from score at the indicated timepoints.
Percentage of Participants Who 'Agree' (Score 5-7) With Each Item (Statement) in the 5 DHEQ Domains at Baseline and Week 24 | Baseline and Week 24
  The DHEQ is a condition-specific measure of OHrQoL in relation to DH. Five DHEQ domains include 34 questions grouped into separate domains: Restrictions, Adaptation, Social Impact, Emotional Impact, and Identity. Participants will score each question using a 7-point scale ranging from 1(strongly disagree) to 7(strongly agree) where lower score indicates better quality of life in relation to DH. Scores 5 to 7 indicates agreement with the statement mentioned in the question, where 5=Agree a little, 6=Agree and 7=Strongly agree. Percentage of participants with scores 5 to 7 for each statement in the 5 DHEQ domains will be reported.
Change From Baseline in Numeric Pain Rating Scale (NPRS) Score at Weeks 1, 2, 4, 8, 12, 16, 20 and 24 | Baseline, Weeks 1, 2, 4, 8, 12, 16, 20 and 24
  NPRS is an 11-point segmented numeric version of a Visual Analogue Scale from which the participant will select a score from 0 to 10 that best reflected the intensity of their pain, where 0=no pain and 10=worst possible pain. Higher score is an indication of greater pain intensity. Change from Baseline will be calculated by subtracting the Baseline score from score at the indicated timepoints.
Satisfaction Numeric Rating Scale (NRS) Score at Week 24 | Week 24
  Participants will be asked to rate their satisfaction with the DH treatment using NRS. NRS is an 11-point ordinal scale used to assess satisfaction with the overall management of the condition for which the participant sought help from treatment. The score ranged from 0 (completely dissatisfied) to 10 (completely satisfied), where higher scores indicate greater satisfaction with DH treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Swathi Varanasi, Principal Investigator — Citruslabs

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.